CLINICAL TRIAL: NCT01917136
Title: Evaluation of Regional Myocardial Perfusion, Glucose Utilization and Oxidative Metabolism in Patients With Pulmonary Hypertension Using Combined [11C]Acetate and [18F]Fluorodeoxyglucose (FDG) PET/CT and Cardiovascular MRI
Brief Title: 11C-acetate/18Fluorodeoxyglucose-FDG PET/CT and Cardiac MRI in Pulmonary Hypertension
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: Brigham and Women's Hospital (Other); University of Maryland (Other); Yale University (Other); Washington University School of Medicine (Other); The Cardiovascular Medical Research and Education Fund (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 817786; NCT01953965 (obsolete NCT alias)
Record Dates: First submitted 2013-08-03; First posted 2013-08-06 (Estimated); Results first posted 2019-02-05 (Actual); Last update posted 2019-02-05 (Actual); Status verified 2018-11

CONDITIONS: Pulmonary Hypertension
Keywords: pulmonary hypertension; right ventricular function; 11C acetate; FDG; ranolazine
MeSH Terms: conditions — Hypertension, Pulmonary | interventions — carbon-11 acetate; Fluorodeoxyglucose F18

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- 11c-acetate and 18F-FDG, and cardiac MRI (Experimental): For each PET/CT imaging session subjects will receive a 15-25 millicurie intravenous injection of 11C-acetate and a 10 millicurie injection of 18F-FDG At baseline/6 months follow up, a cardiac MRI will be performed.
  Interventions: Drug: 11C-acetate; Drug: [18F]Fluoro-2-deoxy-2-D-glucose; Other: Cardiac MRI

INTERVENTIONS:
Drug: 11C-acetate — For each PET/CT imaging session subjects will receive a 15-25 millicurie intravenous injection of 11C-acetate
Drug: [18F]Fluoro-2-deoxy-2-D-glucose — For each PET/CT imaging session subjects will receive a 10 millicurie injection of 18F-FDG
  Other Names: 18F-FDG
Other: Cardiac MRI — Cardiac MRI is performed at 6 months to measure any change in structure and function of the treatment groups.

SUMMARY:
This study is looking at differences in metabolism and functional imaging between pulmonary hypertension subjects with normal right ventricular function and persistent right ventricular dysfunction.

DETAILED DESCRIPTION:
We will measure right ventricular metabolic and structural changes using serial 11C-acetate and 18F-FDG PET/CT and cardiac MRI as response to treatment with ranolazine. Subjects undergo imaging procedures at week 0 and week 26 (optional for normal function patients). This is a companion imaging trial for patients who are eligible for the treatment trial entitled "A randomized, double-blind, placebo controlled, multi-center study to assess the effect of ranolazine on outcomes in subjects with pulmonary hypertension and right ventricular dysfunction accompanied by a comparative study of cellular metabolism in subjects with pulmonary hypertension with and without right ventricular dysfunction". Subjects must enroll in companion treatment protocol to qualify for the imaging protocol.

The cardiac MRI portion of the study continued, but the PET portion of the study was discontinued due to funding.

The treatment protocol is registered under: NCT01839110. Due to funding issues, the completed study was registered under NCT02829034.

ELIGIBILITY:
Inclusion Criteria:

Participation in the companion treatment protocol "A randomized, double-blind, placebo controlled, multi-center study to assess the effect of ranolazine on outcomes in subjects with pulmonary hypertension and right ventricular dysfunction accompanied by a comparative study of cellular metabolism in subjects with pulmonary hypertension with and without right ventricular dysfunction"

Exclusion Criteria:

* Pregnancy or lactation: Women of childbearing potential must have a negative urine or blood pregnancy test on the day of the PET/CT scan.
* Severe anxiety or claustrophobia prohibiting completion of imaging
* Inability to tolerate imaging procedures (1 hour MRI, 30 min and 15 min PET)
* Implantable cardioverter-defibrillator, Pacemaker, hazardous metallic implants or any other contraindication to MRI.
* Uncontrolled diabetes mellitus with fasting glucose > 150 mg/dL

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2013-08 (Actual); Primary Completion 2018-10 (Actual); Study Completion 2018-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yuchi Han, MD, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided
Data available upon request

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 11c-acetate and 18F-FDG, and Cardiac MRI
Started | 21
Completed | 21
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | 11c-acetate and 18F-FDG, and Cardiac MRI
Number analyzed (Participants) | 21
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.4 (15.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 8
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 21

OUTCOME MEASURES:

1. Primary Outcome: Changes in RV Function
Description: RV function as measured by cardiac MRI
Time Frame: 6 months
Population: Patient completed the cardiac MRI at 6 months, changes in RVEF
Measure: Least Squares Mean (Standard Error); unit: percentage
Arm/Group | 11c-acetate and 18F-FDG, and Cardiac MRI
Number analyzed (Participants) | 21
percentage | 7.56 (1.72)

ADVERSE EVENTS:
Time Frame: 7 months
Arm/Group | 11c-acetate and 18F-FDG, and Cardiac MRI
All-Cause Mortality (participants affected / at risk) | 0/21
Serious Adverse Events (participants affected / at risk) | 0/21
Other Adverse Events (participants affected / at risk) | 0/21

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-04-11): https://cdn.clinicaltrials.gov/large-docs/36/NCT01917136/Prot_SAP_000.pdf